CLINICAL TRIAL: NCT07322562
Title: Effects of Music Therapy on Anesthetic Requirements and Hemodynamic Parameters in Thoracic Surgery Patients
Brief Title: Effects of Music Therapy on Anesthetic Requirements and Hemodynamic Parameters
Status: Recruiting | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, mediha turktan, principal investigator, Cukurova University
Other Study IDs: music01
Record Dates: First submitted 2025-12-15; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Hemodynamic Changes; Music Therapy; Thoracic Surgery; Anesthetic Consumption

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Sufi music group: In the sufi music group, sufi music was played through over-ear headphones; the volume was adjusted based on patient comfort and confirmed with the patient. Music playback was initiated alongside routine monitoring and continued throughout the surgery, ending when the patient was transferred to the stretcher after extubation.
  Interventions: Other: music therapy during surgery
- Group 2: Classical Western music group: In the classical Western music group, music was played through over-ear headphones; the volume was adjusted based on patient comfort and confirmed with the patient. Music playback was initiated alongside routine monitoring and continued throughout the surgery, ending when the patient was transferred to the stretcher after extubation.
  Interventions: Other: music therapy during surgery
- Group 3: no music group: In the no music group, the patient was not allowed to listen to any type of music during surgery.

INTERVENTIONS:
Other: music therapy during surgery — In the music groups, music was played through over-ear headphones; the volume was adjusted based on patient comfort and confirmed with the patient. Music playback was initiated alongside routine monitoring and continued throughout the surgery, ending when the patient was transferred to the stretcher after extubation. For infection control purposes, headphone sponges were changed for each patient.
  Groups: Group 1: Sufi music group; Group 2: Classical Western music group

SUMMARY:
Music therapy has been reported to reduce analgesic and anesthetic requirements, but evidence in thoracic surgery remains limited. This prospective observational study aimed to evaluate the effects of different music types on hemodynamic stability and anesthetic consumption in patients undergoing thoracic surgery.

DETAILED DESCRIPTION:
After institutional ethics approval and written informed consent, 159 adult patients (ASA I-III) scheduled for elective thoracic surgery under general anesthesia were enrolled. Patients were randomized by sealed-envelope method into three groups: Group T (Sufi music), Group B (Classical Western music), and Group C (control, no music). Music was delivered via over-ear headphones from induction until the end of surgery. Sedation was evaluated using the Riker Sedation-Agitation Scale (RSAS), and pain using the Visual Analog Scale (VAS). Hemodynamic variables, anesthetic agent consumption, and postoperative recovery parameters were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over,
* American Society of Anesthesiologists (ASA) classification I-III,
* No hearing acuity,
* Volunteer to participate in the study,
* Cooperative and oriented,
* No history of psychiatric illness and/or psychiatric medication use,

Exclusion Criteria:

* Patients who were under 18 years,
* ASA classification >III,
* had hearing loss,
* had a psychiatric diagnosis and/or were taking antipsychotic/antidepressant/mood stabilizer medications,
* were uncooperative (dementia, mental retardation, etc.),
* Major complications during the intraoperative or postoperative period, (respiratory failure, hemodynamic instability, hypoxia, serious arrhythmia, cardiac arrest, etc.)
* Emergency surgery,
* had a history of alcohol or drug abuse,
* did not speak Turkish,
* did not consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who will undergo thoracic surgery under general anesthesia and meet the criteria of being over 18 years of age
Sampling Method: Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
anesthetic consumption | during surgery
  desfluran consumption during surgery (mL)
anesthetic consumption | during induction of anesthesia
  Induction propofol dose (mg)

SECONDARY OUTCOMES:
hemodynamic parameters | during surgery, 48 hour after surgery
  systolic blood pressure (mmHg)
hemodynamic parameters | during surgery, 48 hour after surgery
  diastolic blood pressure (mmHg)
hemodynamic parameters | during surgery, 48 hour after surgery
  mean arterial pressure (mmHg)
hemodynamic parameters | during surgery, 48 hour after surgery
  heart rate (beats/min)

CONTACTS AND LOCATIONS:
Overall Officials: Mediha Turktan, M.D., Principal Investigator — Cukurova University
Locations (1):
- Cukurova University Faculty of Medicine Anesthesiology Department, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No